CLINICAL TRIAL: NCT04568551
Title: COVID-19-associated Anxiety of Pregnant Women for Anomalies, Stillbirth and Preterm Labor - CAASPtrial
Brief Title: COVID-19-associated Anxiety of Pregnant Women for Anomalies, Stillbirth and Preterm Labor
Acronym: CAASP
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Marcus Riemer, MD, Dr. med. Marcus Riemer, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKGEB001
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Capture of anxiety for anomalies, stillbirth and preterm Labor of pregnant women during COVID-19 pandemia

ELIGIBILITY:
Inclusion Criteria:

* consenting ability

Exclusion Criteria:

* language barrier
* uncompleted questionary

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women between 33 until 37 weeks of Gestations with planned Labor in University Hospital of Halle or St.Elisabeth and St.Barbara Hospital Halle, Germany
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
anxiety for anomalies during COVID-19-pandemic and before (percentage difference in agreement to the items of the questionnaire) | 6 months
  Measurement of self-reported anxiety by a questionnaire and State-Trait Anxiety Inventory (STAI) and comparison with different empiric studies of anxiety for anomalies in pandemics
anxiety for stillbirths during COVID-19-pandemic and before (percentage difference in agreement to the items of the questionnaire) | 6 months
  Measurement of self-reported anxiety by a questionnaire and State-Trait Anxiety Inventory (STAI) and comparison with different empiric studies of anxiety for stillbirths in pandemics
anxiety for preterm labour during COVID-19-pandemic and before (percentage difference in agreement to the items of the questionnaire) | 6 months
  Measurement of self-reported anxiety by a questionnaire and State-Trait Anxiety Inventory (STAI) and comparison with different empiric studies of anxiety for preterm labour in pandemics

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Halle, Halle, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: Undecided